CLINICAL TRIAL: NCT01285570
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Intravenous (IV) Ulimorelin Administered Post-Operatively to Accelerate Recovery of Gastrointestinal (GI) Motility in Subjects Who Have Undergone Partial Bowel Resection
Brief Title: Ulimorelin Study of Efficacy and Safety (ULISES 007)
Acronym: ULISES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tranzyme, Inc. (Industry)
Collaborators: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TZP-101-CL-P007
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Gastrointestinal Dysmotility
MeSH Terms: interventions — Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Experimental 2 (Experimental)
  Interventions: Drug: Ulimorelin Intravenously (IV)
- experimental 1 (Experimental)
  Interventions: Drug: Ulimorelin Intravenously (IV)
- Placebo (Placebo Comparator): Placebo comparator daily (QD)
  Interventions: Drug: 5% dextrose in water

INTERVENTIONS:
Drug: Ulimorelin Intravenously (IV) — 480 microg/kg daily (QD)
  Arms: Experimental 2
Drug: Ulimorelin Intravenously (IV) — 160 microg/kg daily (QD)
  Arms: experimental 1
Drug: 5% dextrose in water — Placebo
  Arms: Placebo

SUMMARY:
Post-operative administration of ulimorelin is expected to reduce time to recovery of Gastrointestinal (GI) function in patients who have undergone partial large bowel resection.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18 to 80 years of age, inclusive
* Scheduled to undergo open bowel resection with colonic anastomosis.
* For women who can potentially become pregnant a pregnancy test at screening and admission must be negative.

Exclusion Criteria:

* Weight more than 200kg (441 pounds)
* Pregnant or breastfeeding
* Known history of drug or alcohol abuse within the previous year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Recovery of GI Function | up to 7 days of dosing or until hospital discharge

SECONDARY OUTCOMES:
Ancillary GI Functions | up to 7 days of dosing or hospital discharge

CONTACTS AND LOCATIONS:
Locations (45):
- United States (23):
  - Fountain Valley Regional Hospital, Fountain Valley, California
  - Orange Coast Memorial Med. Ctr., Fountain Valley, California
  - USC, Colorectal Surgery Division, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Denver VA Medical Center, Denver, Colorado
  - Nature Coast Clinical Research, Inverness, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Pensacola Research Consultants, Pensacola, Florida
  - Sunrise Clinical Research, Inc., Sunrise, Florida
  - ARS Clinical Trials, Powder Springs, Georgia
  - So. Illinois Univ. School of Medicine, Springfield, Illinois
  - Univ. of Louisville, Dept. of Surgery, Louisville, Kentucky
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - CRC of Jackson, Jackson, Mississippi
  - Creighton Univ. Medical Ctr., Omaha, Nebraska
  - Mt. Sinai Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Case Medical Ctr., Cleveland, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - Mt. Talbert Medical Offices, Clackamas, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - JPS Health Network, Dept. of Surgery, Fort Worth, Texas
  - Southwest Surgical Associates, Houston, Texas
- Hungary (4):
  - JohnFerenc Del-pesti Hospital, Budapest
  - Petz Aladar County Education Hospital, Győr
  - County Hospital of Kecskemet, Kecskemét
  - St. Gyorgy Hospital of Fejer County, Székesfehérvár
- Italy (3):
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - Policlinico Universitario Agostino Gemelli -Univ, Rome
  - IRCCS Policlinico San Donato, San Donato
- Poland (3):
  - Plac Hallera, Genl Surgery, Lodz
  - Univ. Hospital #1, N. Barlicki Med. Univ., Lodz
  - Hospital Wolski, Warsaw
- Romania (5):
  - Spitalul Clinic de Urgenta "Prof. Dr. Octavian Fodor", Cluj-Napoca
  - Spitalul Clinic Judetean de Urgente, Iași
  - Spitalul Clinic Judetean de Urgenta Oradea, Oradea
  - Spitalul Clinic Judetean Mures, Târgu Mureş
  - Spitalul Clinic Judetean de Urgenta Timisoara, Timișoara
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Bezanijska Kosa, Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - Clinical Center Nis, Niš
- United Kingdom (3):
  - Nottingham University Hospital, Nottingham
  - Scarborough Hospital, Scarborough
  - Northern General Hospital, Sheffield

REFERENCES:
- [Derived] Shaw M, Pediconi C, McVey D, Mondou E, Quinn J, Chamblin B, Rousseau F. Safety and efficacy of ulimorelin administered postoperatively to accelerate recovery of gastrointestinal motility following partial bowel resection: results of two randomized, placebo-controlled phase 3 trials. Dis Colon Rectum. 2013 Jul;56(7):888-97. doi: 10.1097/DCR.0b013e31829196d0. PMID 23739196